CLINICAL TRIAL: NCT05403346
Title: Clinical Evaluation of a SARS-CoV-2 CoviDx™COVID-19 Antigen Self-Test
Brief Title: Clinical Evaluation of a COVID-19 Antigen Self-Test (CoviDx™)
Acronym: CoviDx™
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to the difficulty to enrol patients
Sponsor: Lumos Diagnostics (Industry)
Collaborators: Rapid Pathogen Screening (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-0010
Record Dates: First submitted 2022-06-01; First posted 2022-06-03 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-06

CONDITIONS: SARS-CoV-2; Covid19
Keywords: Antigen; Rapid Point of care testing; Self testing
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mid turbinate nasal swabs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SARS COv-2 RT-PCR AND Self collected CoviDx Covid-19 Antigen Self-Test: Sequentially enrolled symptomatic patients will have a nasal swab collected for high-sensitive SARS-CoV-2 RT-PCR testing as comparator and self collect a nasal swab for CoviDx™ Covid-19 Antigen self-testing. Order of tests will be performed following a randomization scheme.
  Interventions: Device: CoviDx™ Covid-19 Antigen Self-Test

INTERVENTIONS:
Device: CoviDx™ Covid-19 Antigen Self-Test — All patients will self-collect a mid-turbinate nasal swab for CoviDx™ Covid-19 Antigen self-testing

SUMMARY:
Prospective study that will evaluate the clinical agreement of the CoviDx™ Self test compared to SARS-CoV-2 RT-PCR.

DETAILED DESCRIPTION:
Subjects who are currently experiencing symptoms associated with COVID-19 will be enrolled. Each enrolled subject will either self-collect one sample from the anterior nares or have the sample collected by another lay individual. Each subject will then have a mid-turbinate nasal swab sample collected for comparator test

ELIGIBILITY:
Inclusion Criteria:

* Mid-turbinate nasal swab collected for SARS-CoV-2 RT-PCR at the same time of CoviDx Rapid Antigen swab collection
* Symptomatic subjects suspected of having COVID-19, first onset of COVID-19-like symptoms (e.g., chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, or diarrhea) should not have started more than 5 days from the time of the study visit. Symptoms must be present on the day of CoviDx testing.
* ≥ 2 years of age
* Participants between 2-13 years of age, inclusive, must participate with a guardian who will be collecting the swab.
* Signed Informed Consent

Exclusion Criteria:

* Participants with prior medical or laboratory training
* Unable or unwilling to provide signed, Informed Consent
* Less than 2 years of age
* Received a positive diagnostic test result for COVID-19 in the past 14 days
* Received a negative diagnostic test result for COVID-19 in the last 18 hours
* Study Comparator collection that occurred > 3 hours from CoviDx swab collection
* For symptomatic participants: first onset of COVID-19-like symptoms occurring more than 5 days from study visit
* Invalid or missing study comparator test results
* Use of a non-high-sensitive SARS-CoV-2 test as the comparator SARS-CoV-2 RT-PCR test (e.g., rapid molecular, rapid antigen tests, tests that do not have FDA EUA, a test that was not approved by Sponsor for use in the study)
* Enrollment in another study involving the collection of a nasopharyngeal, mid-turbinate nasal swab or anterior nasal swab within 6 hours of CoviDx testing.
* Indicates they would not use a COVID-19 diagnostic test kit in real life
* Taking any of the following medications or treatments within 7 days of study visit (antivirals (e.g., Remdesivir, Paxlovid) and/or monoclonal antibodies (e.g., REGEN-COV (casirivimab, imdevimab), Sotrovimab (Xevudy), Evusheld)
* Nasal spray administration in the last 48 hours

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lay users who do not have medical or laboratory experience significant experience performing repeated self-testing. Subjects will be 2 years of age or older and have symptoms of COVID-19 that started ≤ 5 days from their study visit
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Performance of CoviDx Covid-19 Antigen Self-Test in nasal swab as compared to a high-sensitive SARSCoV- 2 RT-PCR granted Emergency Use Authorization (EUA) by the FDA | 60 days
  Evaluate the performance (positive percent agreement (PPA) and negative percent agreement (NPA)) of the CoviDx™ COVID-19 Antigen Self-Test for the detection of SARS-CoV-2 virus antigen in anterior nasal swab (NS) samples collected by lay users compared to results obtained from by a high-sensitive SARS-CoV-2 RT-PCR granted Emergency Use Authorization (EUA) by the FDA (comparator test).

CONTACTS AND LOCATIONS:
Locations (1):
- PAS Research, Tampa, Florida, United States